CLINICAL TRIAL: NCT01781689
Title: The Relationship Between Motor Cortex Oxygenation and Motor Function Recovery in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Zheng-Yu Hoe, MD., PhD., Principal Investigator, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: VGHKS102-086; VGHKS12-CT7-07 (Other: Kaohsiung V.G.H. Institutional Review Board)
Record Dates: First submitted 2013-01-27; First posted 2013-02-01 (Estimated); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Stroke
Keywords: cortical activation; motor function; activity of daily living
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Functional Electric Stimulation (Experimental): perform arm cranking with functional electrical stimulation
  Interventions: Procedure: Functional Electric Stimulation
- traditional rehabilitation program (Sham Comparator): Receive traditional rehabilitation programs
  Interventions: Other: Rehabilitation programs
- Health (No Intervention): with no motor function impairment

INTERVENTIONS:
Procedure: Functional Electric Stimulation — apply to the hemiplegia affected limbs, helping movement
  Arms: Functional Electric Stimulation
Other: Rehabilitation programs — include occupational therapy and physical therapy
  Arms: traditional rehabilitation program

SUMMARY:
Stroke is the most common cause of motor function impairment. However, the functional impairment is not totally irreversible. Several mechanisms may involved in both the cortical and motor function recovery after onset of stroke, and most of them are related to changes of cortical perfusion and metabolism.

Motor function recovery after stroke (especially middle cerebral artery territory lesion) frequently follow stereotypic pattern (brunnström stage).

This study is designed to investigate the relationship between motor cortex oxygenation/metabolism and motor function recovery after stroke. To seek if there is similar stereotypic pattern of motor cortex oxygenation/metabolism change during the recover stage after stroke.

DETAILED DESCRIPTION:
Participants receive evaluations (1/week for 3 months period) of

* motor function (Include: MMSE, brunnström stage, Fugl-Meyer Assessment of Physical Performance, Box and Block Test of Manual Dexterity, Functional Independence Measure)
* cortical perfusion detection during performing limb movements (using NIRS)

Then use path analysis to investigate the relationship between motor cortex oxygenation/metabolism and motor function recovery after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke(unilateral, onset within 7 days, without previous stroke history)
* Vital sign stable
* Upper extremity motor function impairment(brunnström stage I~III)

Exclusion Criteria:

* with pacemakers
* Seizure history
* Serious dysrhythmias
* Poor cognition function(MMSE<13)

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-10; Primary Completion 2019-07-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Cortical activation | weekly changes within 3 months
  Using Near-infrared spectroscopy to measure cortical activation changes weekly for 3 months

SECONDARY OUTCOMES:
motor function | weekly changes within 3 months
  assess motor function every week for 3 months

OTHER OUTCOMES:
Activity of daily living function | weekly changes within 3 months
  assess Activity of daily living function weekly for 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Zheng-Yu Hoe, Principal Investigator — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan